CLINICAL TRIAL: NCT03650257
Title: A Large-scale Research for Immunotherapy of Glioblastoma With Autologous Heat Shock Protein gp96
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cure&Sure Biotech Co., LTD (Industry)
Collaborators: Beijing Tiantan Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-TT-G-02
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Glioma of Brain
Keywords: supratentorial glioma
MeSH Terms: interventions — glucose-regulated proteins; Heat-Shock Response; vitespin; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- gp96 group (Experimental): Patients receive standard treatment with radiation and temozolomide after surgery.
  Then 6 times of autologous gp96 vaccination are administered via subcutaneous injection in 25μg doses at the 2nd week after the end of postoperative radiotherapy.
  ( gp96 is administered once a week for the first 4 weeks, the 5th injection is administered 2 weeks after the 4th injection, and the 6th injection is administered 3 weeks after the 5th injection. )
  The first adjunctive temozolomide startes on the day of the fifth gp96 injection.
  (150-200 mg/m2/day for 5 days, then stop for 23 days, one cycle is 28 days for a total of 6 cycles)
  Interventions: Biological: gp96; Drug: Temozolomide; Radiation: radiotherapy
- control group (Active Comparator): Patients receive standard treatment with radiation and temozolomide after surgery. Then only adjuvant treatment with temozolomide is administered.
  Interventions: Drug: Temozolomide; Radiation: radiotherapy

INTERVENTIONS:
Biological: gp96 — 25 mcg IH
  Other Names: Heat Shock; HSPPC-96
  Arms: gp96 group
Drug: Temozolomide — temozolomide monotherapy (150-200 mg / m2 / day for 5 days, then discontinuance for 23 days , 28 days for a a cycle, a total of 6 cycles ).
  Other Names: TZM
Radiation: radiotherapy — Stupp regimen of radiotherapy

SUMMARY:
This trial is to further study the safety and effectiveness of autologous gp96 treatment of glioblastoma on the basis of preliminary work.

DETAILED DESCRIPTION:
RATIONALE: heat shock protein gp96-peptide complex made from a person's tumor cells may help the body build an effective immune response to kill tumor cells.

Overall Goals:

- to evaluate the safety and induction of anti-tumor immunity by administration of an immunogenic human tumor cell vaccine, and assess immune response in relation to clinical outcome.

Primary Aim:

- to further evaluate effectiveness of autologous gp96 treatment of glioblastoma on the basis of preliminary work.

Secondary Aims:

to study the immune response to vaccination, to monitor clinical responses , to further the safety of vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the informed consent document; must sign the informed consent;
2. Aged 18 to 75 years old , sex is not limited;
3. Newly Diagnosed supratentoria glioma, Must have undergone a at least a 80% resection;
4. Availability of at least 4 g tumor sample;
5. Patient must receive concurrent chemoradiotherapy (temozolomide chemotherapy and radiotherapy).
6. Karnofsky functional status rating > or equal to 70.
7. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; Hemoglobin > 10g/dL ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], alanine amino transferase [ALT] <2.5 times institutional upper limit of normals [IULNs] ), and adequate renal function (BUN and creatinine <1.5 times IULNs)
8. Agree to Surgical indications of Heart & lung and without the coagulation system disease
9. Except for surgery and radiotherapy and chemotherapy before vaccine treatment, no other cancer treatment is received.

Exclusion Criteria:

1. Inability to comply with study-related procedures
2. Unavailability of at least 6 doses of vaccine
3. Severe allergies
4. Unstable or severe intercurrent medical conditions
5. Current diagnosis of Human Immunodeficiency Virus and Patients with active uncontrolled infection.
6. patients with any systemic disease needed to be treated with immunosuppressant or Corticosteroids.
7. any other clinical trials within 30 days pre-vaccination.
8. Female patients who are pregnant or breastfeeding
9. Carmustine extended release implant surgery within 6 months
10. Steroidal drugs are currently being used systemically.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | 1 years

SECONDARY OUTCOMES:
Progression-free survival rate | 1 year
Progression-free survival | 5 years
Overall survival | 5 years
changes in antigen specific T cells | within 3 days before the first vaccination and within 10 days after the last vaccination
  tumor antigen specific T cells are determined by IFN-γ Enzyme-linked Tumor antigen specific T cells will be determined by IFN-γ Enzyme-linked immunosorbent spot using the autologous tumor cell lysis as the antigen.
Number of participants with adverse events related to gp96 immunotherapy | up to 3 months after vaccine completion
  A complete blood count will be requested before the first vaccination, after the second vaccination and after the last vaccination to monitor the side effect of gp96 immunotherapy. And blood chemistries will also be requested at the same time point for the same reason.And other adverse events related to gp96 immunotherapy will be recorded according to the NCI-CTCAE 5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: zhixian Gao, Doctor, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China